CLINICAL TRIAL: NCT04955873
Title: Ridge Preservation With the Use of a Xenogenic Bone Graft Material (Symbios Xenograft Granules) and a Pre-hydrated Collagen Membrane Symbios Pre-hydrated Collagen Resorbable Membrane): A Pilot Multicenter Randomized Controlled Study
Brief Title: Ridge Preservation Using Xenogenic Bone Graft and Pre-hydrated Collagen Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Bruno Kessler (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-BI-16-004
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Alveolar Bone Resorption; Edentulous Alveolar Ridge
Keywords: Ridge preservation; Xenograft; Collagen membrane; Socket preservation; Socket management; Biomaterial; Histomorphometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test - Group A - Dentsply biomaterials (Experimental): Dental extraction socket treated with the combined use of the xenogenic bone granules "Dentsply Sirona Symbios Xenograft Granules" and the resorbable collagen membrane "Dentsply Sirona Symbios Collagen Membrane SR".
  Interventions: Device: Treatment of the dental extraction socket using newly-released biomaterials
- Active comparator - Group B - Geistlich biomaterials (Active Comparator): Dental extraction socket treated with the combined use of the xenogenic bone granules "Geistlich Bio-oss Collagen" and the resorbable collagen membrane "Geistlich BioGide".
  Interventions: Device: Treatment of the dental extraction socket using well-known biomaterials
- Control - Group C - Spontaneous healing (No Intervention): Spontaneous postextraction alveolar healing

INTERVENTIONS:
Device: Treatment of the dental extraction socket using newly-released biomaterials — Treatment of the dental extraction socket with the combined use with the combined use of a newly-released xenogenic bone granules and a resorbable collagen membrane.
  Arms: Test - Group A - Dentsply biomaterials
Device: Treatment of the dental extraction socket using well-known biomaterials — Treatment of the dental extraction socket with the combined use of a well-known xenogenic bone granules and a resorbable collagen membrane
  Arms: Active comparator - Group B - Geistlich biomaterials

SUMMARY:
This pilot multicentric randomized controlled clinical trial is aimed at evaluating the composition of the new-formed tissue into the dental socket after 6 months from tooth extraction and the application of a combination of xenograft bone granules and collagen membrane. Extraction sites will be either grafted with Dentsply Symbios Xenograft Granules and covered with Dentsply Symbios pre-hydrated Collagen Resorbable Membrane or grafted with Geistlich Bio-Oss Collagen and covered with Geistlich Bio-Gide membrane. Results will be compared to spontaneous socket healing.

DETAILED DESCRIPTION:
Rational

Socket preservation techniques are effective in mitigating the dimensional changes of the alveolar socket that spontaneously occur after tooth extraction (Avila-Ortiz G, et al. 2019). However, there is insufficient information regarding the type and quality of the newly formed tissue at the extraction site before implant positioning.

Study design

This study is a three-arm multicentric randomized trial that will evaluate the bone healing following ridge preservation of extraction sockets using two different combinations of commercially available xenograft bone granules and collagen membranes available in the market. Results will be compared to tissues obtained from spontaneous healing. A total of 45 participants (15 in each arm) is expected.

Study protocol

Patients, satisfying inclusion criteria and having signed study informed consent, will be randomly allocated to three study groups, receiving the following treatments at the time of tooth extraction:

* Group A: grafting of postextraction socket with Dentsply Symbios Xenograft granules covered with Dentsply Symbios pre-hydrated Collagen Resorbable Membrane (Test - Group A)
* Group B: grafting of postextraction socket with Geistlich Bio-Oss Collagen and covering with Geistlich Bio-Gide Collagen membrane (Active comparator - Group B)
* Group C: no further treatment of the postextraction socket (spontaneous healing, Control - Group C) After 6 months from the extraction, radiographic examinations will be performed and the implant surgery will take place.

On the day of the surgery the width of keratinized mucosa at socked site will be registered. Then, following loco-regional anesthesia, a soft tissue sample of 3 mm in diameter will be obtained using a circular punch at the site intended to receive the implant. Subsequently, a flap will be elevated. Using a trephine drill a 3 mm in diameter block of hard tissue with a length of 5- 6 mm will be collected. The preparation of the implant site will be then carried out until the desired diameter and length are reached for the insertion of the corresponding implant. Torque at implant insertion will be registered.

Once the implant has been inserted, the healing abutment will be positioned and soft tissues will be sutured with single sutures. The prosthetic rehabilitation will be completed after osseointegration, approximately 3 months after the implant surgery.

Histological analysis of soft tissue and hard tissue biopsies

Tissue samples will be immediately fixed in formalin after collection. Histological analysis will be performed on formalin-fixed paraffin-embedded tissue sections, to determine the quantity and quality newly formed tissue and the remaining fraction of the implanted biomaterials.

More specifically, the collected tissue biopsies will be fixed in 4% buffered formalin, decalcified into ethylenediaminetetraacetic acid (EDTA) (if necessary), dehydrated and included in paraffin. Serial sections, including the central portion of the biopsy, will be prepared and colored in hematoxylin and eosin. Vascular structures will be identified by CD34 (Cluster of differentiation 34, hematopoietic progenitor cell antigen) antibody. Portions occupied by mineralized bone (lamellar bone, trabecular bone), osteoid (partially mineralized connective tissue matrix rich in collagen), bone marrow (adipocytes and vascular structures), fibrous tissue (unorganized collagen fibers, cells and vessels), biomaterial granules and residual tissue (unidentified tissue elements, preparation artifacts) will be characterized by morphometric measurements performed according to the protocol described by Lindhe et al. (Clin. Oral Impl. Res.2014;25:786-790). Soft tissues characterization will include the analysis of the structural composition of epithelial and connective tissues, the quantification of the amount micro-vessels in connective tissue, the definition of the inflammatory cell types, and the collagen tissue content according to protocols described in Tomasi et al. (J Clin Periodontol. 2016;43:816-24).

Data analysis and statistics

Data analysis will be aimed at detecting statistically significant differences in tissue composition between the group A in respect to the most appropriate of the two remaining groups (e.g. the percentage of bone tissue in the test group will be compared with that of control group C while the percentage of residual biomaterial six months after implantation will be compared with the active control B). Statistically significant differences with p<0.05 will be considered.

Data normality will be verified with the Shapiro-Wilk test. Outcome variables for each of three groups will be expressed by means of mean ± standard deviation for continuous variables with normal distribution, or by means of median and value at the 25th and 75th percentile for variables with non-normal distribution. Parametric or non-parametric statistical tests will then be applied to compare between groups, according to data normality.

ELIGIBILITY:
Inclusion Criteria:

* have at least one tooth (from the central incisor to the second permanent molar) to be extracted and replaced with an endosseous implant;
* no need of a temporary prosthesis;
* availability to participate to the follow-up;
* sign the study informed consent and consent to data treatment;

Exclusion Criteria:

* less than 20 years;
* known allergy to collagen or bone graft material;
* contraindications to implant therapy;
* ongoing bisphosphonate-based therapy;
* ongoing high-dose corticosteroid therapy;
* relevant co-morbidities of the maxillary bones that interfere with bone remodeling (degenerative bone diseases, osteomyelitis at the extraction site or surrounding areas, subacute mandibular osteitis, local microvascular disorders);
* smoking;
* pregnancy;
* metabolic diseases (diabetes, hyperparathyroidism);
* systemic bone diseases;

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Composition of new-formed hard tissue into the post-extractive socket | Six months after surgery
  Amount of mineralized bone, residual biomaterial, fibrous tissue
Composition of new-formed soft tissue over the post-extractive socket | Six months after surgery
  Amount of epithelial tissue, connective tissue, of neovascularization, inflammatory cells, residual collagenic biomaterial

SECONDARY OUTCOMES:
Implant torque at insertion | Six months after surgery, at implant insertion.
  Dynamometric measurement of the insertion torque at implant placement
Width of keratinized mucosa | Six months after surgery, at implant insertion.
  Extension of keratinized mucosa in the bucco-lingual direction

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Tessarolo, PhD, Principal Investigator — Bruno Kessler Fundation, Trento Italy; Paolo Ghensi, DDS, PhD, Principal Investigator — Università degli Studi di Trento
Locations (5):
- Italy (5):
  - Studio Odontoiatrico Maia Dentis, Merano, Bolzano
  - Studio Medico Dentistico Dott. Mandelli, Pioltello, Milano
  - Studio Dentistico Bressan Associati Di Bressan Eriberto - Bressan Giuseppe - Bressan Paolo, Chions, Pordenone
  - Studio Dentistico Associato Tomasi-Ghensi-Varotto, Cembra, Trento
  - Studio Dentistico Donati Di Donati Andrea & Mauro, Perugia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Lindhe J, Cecchinato D, Donati M, Tomasi C, Liljenberg B. Ridge preservation with the use of deproteinized bovine bone mineral. Clin Oral Implants Res. 2014 Jul;25(7):786-90. doi: 10.1111/clr.12170. Epub 2013 Apr 4. PMID 23556467
- [Background] Tomasi C, Tessarolo F, Caola I, Piccoli F, Wennstrom JL, Nollo G, Berglundh T. Early healing of peri-implant mucosa in man. J Clin Periodontol. 2016 Oct;43(10):816-24. doi: 10.1111/jcpe.12591. Epub 2016 Jul 28. PMID 27329966